CLINICAL TRIAL: NCT02021344
Title: Mental Health First Aid for College Students: A Multi-campus Randomized Control Trial of a Community Health Intervention
Brief Title: Mental Health First Aid for College Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Daniel Eisenberg, Associate Professor, Department of Health Management & Policy, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: NIMH 1RC1MH089757-01; 1RC1MH089757-01 (NIH)
Record Dates: First submitted 2013-12-14; First posted 2013-12-27 (Estimated); Last update posted 2013-12-27 (Estimated); Status verified 2013-12

CONDITIONS: Depression; Anxiety; Suicidal Ideation; Eating Disorders
MeSH Terms: conditions — Depression; Anxiety Disorders; Suicidal Ideation; Feeding and Eating Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Pure control (No Intervention): Practice as usual (no MHFA) in all residences on these campuses.
- Intervention residence on mixed campus (Experimental): Mental Health First Aid delivered to these residences, but not all other residences at the same campus.
  Interventions: Behavioral: Mental Health First Aid
- Pure intervention residence (Experimental): Mental Health First Aid delivered to this residence and all other residences at the same campus
  Interventions: Behavioral: Mental Health First Aid
- Control at mixed campus (No Intervention): Practice as usual (no MHFA) at this residence, but some other residences at same campus are in experimental condition (MHFA).

INTERVENTIONS:
Behavioral: Mental Health First Aid — Originally developed in 2001, MHFA is a 12-hour course comprised of six modules, covering depression, anxiety, psychosis, substance abuse, eating disorders, and self-harm. Each module includes information about the mental health-related problems (e.g., signs and symptoms), advice on how to respond appropriately, and interactive activities to enhance the learning process. Some modules include videos with perspectives of individuals recovering from mental disorders and examples of how to effectively use the MHFA intervention. Program participants learn how to help individuals in crisis and also how to recognize early warning signs and intervene before mental health problems progress to crises.
  Arms: Intervention residence on mixed campus; Pure intervention residence

SUMMARY:
Most college students with mental disorders do not receive treatment, and over 80% of those who die by suicide have never made contact with campus mental health services. Knowledge, stigma, and other health beliefs represent significant barriers to help-seeking for many of these students. However, there have been no large-scale intervention studies for reducing these barriers to mental health treatment on college campuses. This project will fill this gap by determining whether a community mental health education program, Mental Health First Aid (MHFA), is an effective method to increase number of students who seek mental health services on college campuses. MHFA is an international, 12-hour training program that has been shown to increase knowledge of mental illnesses and their treatments, decrease stigma, and increase helping behaviors in community members. However, it has not been tested in a college setting in the United States. To determine the effectiveness of MHFA in US colleges, the proposed project will involve a randomized control trial of the MHFA training program on 32 campuses representing a range of higher education institutions, from community colleges in rural areas to research universities in large, urban areas. The MHFA training program will be administered to peer supports such as residential advisors. Administrative data from campus mental health services and pre- and post-intervention surveys will be used to collect outcome data on service utilization, knowledge, attitudes, and other measures. Data analyses will focus on identifying changes in students' behaviors, knowledge, and attitudes toward mental illnesses that can be attributed to the MHFA training. In addition to testing a novel and timely mental health intervention for college students, this project will result in improved data collection measures for college populations, and will lay the foundation for stronger connections and future collaborations between diverse campus communities. If the MHFA program is successful in reducing stigma and increasing general on-campus awareness and early treatment of emerging mental health problems, then it may provide a cost-effective means for enabling more students to seek early treatments for developing mental health problems.

ELIGIBILITY:
Inclusion Criteria:

* Student enrolled in a participating campus as a full-time, residential undergraduate during the 2009-2010 or 2010-2011 academic years. Student must have been living in a participating residence hall.

Exclusion Criteria:

* Students under 18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2543 (Actual)
Dates: Start 2009-09; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Changes in mental health service utilization | baseline, 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Eisenberg, PhD, Principal Investigator — University of Michigan; Nicole L Speer, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] Richardson R, Dale HE, Robertson L, Meader N, Wellby G, McMillan D, Churchill R. Mental Health First Aid as a tool for improving mental health and well-being. Cochrane Database Syst Rev. 2023 Aug 22;8(8):CD013127. doi: 10.1002/14651858.CD013127.pub2. PMID 37606172